CLINICAL TRIAL: NCT00731562
Title: Phase 1, Open-Label, Randomized, Single-Dose, Two-Way Crossover Study To Evaluate The Effect Of Food On The Oral Bioavailability Of A Varenicline Controlled Release Formulation In Healthy Adult Smokers
Brief Title: An Investigation Of The Effects Of Food On The Absorption Of A Varenicline Controlled Release Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A3051088
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Pharmacokinetics; Bioavailability; Smoking Cessation
Keywords: food, varenicline, pharmacokinetics, bioavailability
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline Controlled Release, Fasted (Experimental)
  Interventions: Drug: Varenicline Tartrate Controlled Release
- Varenicline Controlled Release, Fed (Experimental)
  Interventions: Drug: Varenicline Tartrate Controlled Release

INTERVENTIONS:
Drug: Varenicline Tartrate Controlled Release — A single, 2.4 mg dose of a varenicline controlled release tablet administered orally under fasted conditions
  Arms: Varenicline Controlled Release, Fasted
Drug: Varenicline Tartrate Controlled Release — A single, 2.4 mg dose of a varenicline controlled release tablet administered orally under fed conditions
  Arms: Varenicline Controlled Release, Fed

SUMMARY:
1. To estimate the absorption of a single oral dose of a controlled release varenicline tablet under fed and fasted conditions.
2. To evaluate the pharmacokinetics, safety, and tolerability of a single dose of a varenicline controlled release tablet under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adult smokers
* 18 to 55 years of age

Exclusion Criteria:

* Sensitivity to varenicline
* Illegal drug use
* Pregnant or nursing females

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Varenicline area under the curve (AUC) from time of study medication administration to last quantifiable plasma concentration (AUClast) and AUC from time of study medication administration to infinity (AUCinf). | 5 days
Maximum plasma concentration of varenicline | 1 day

SECONDARY OUTCOMES:
Safety measures including adverse events | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, East Grand Forks, Minnesota
  - Pfizer Investigational Site, Fargo, North Dakota

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051088&StudyName=An%20Investigation%20Of%20The%20Effects%20Of%20Food%20On%20The%20Absorption%20Of%20A%20Varenicline%20Controlled%20Release%20Formulation